CLINICAL TRIAL: NCT04628169
Title: Impact of Netrin-1 in the Pathophysiology of Placenta Accreta Spectrum
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hanaa Mohammed Mohammed Sayed, assistant lecturer, Assiut University
Other Study IDs: netrin-1 in placenta accreta
Record Dates: First submitted 2020-11-09; First posted 2020-11-13 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Pathophysiology of Placenta Accreta
Keywords: Netrin-1, neogenin,PAS, zeb-1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: 30 placental specimens of PAS
  Interventions: Other: no intervention applied
- group B: 30 placental specimens of heaithy women with normal pregnancy
  Interventions: Other: no intervention applied

INTERVENTIONS:
Other: no intervention applied — no intervention applied

SUMMARY:
The main goal of this study is to assess the role of Netrin 1, neogenin and ZEB1 in PAS-associated invasion

DETAILED DESCRIPTION:
* To evaluate the immunohistochemical expression of these proteins in PAS specimens in comparison with the control placental tissues.
* To correlate their expression with the demographic parameters.
* To assess the correlation between their expression in PAS specimens.

ELIGIBILITY:
inclusion criteria

* PAS patients who underwent hysterectomy to allow proper pathologic grading of PAS

exclusion criteria

* patients with fundal and middle anterior or posterior placenta,
* pregnancy associated with morbid conditions such as hypertension, diabetes mellitus, autoimmune disease, cardiac disease, renal disease, history of anemia, blood transfusion, other blood diseases and endocrinal disease; fetal distress or intrauterine growth retardation.
* uterine scar pregnancies were excluded

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: 30 PAS specimens and 30 placental specimens from matched control.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
impact of netrin-1 in the pathophysiology of placenta accreta spectrum | baseline
  1. Evaluation of the immunohistochemical expression of netrin 1 in PAS specimens in comparison with the control placental tissues.
  2. Evaluation of the immunohistochemical expression of neogenin in PAS specimens in comparison with the control placental tissues
  3. Evaluation of the immunohistochemical expression of ZEB1 in PAS specimens in comparison with the control placental tissues.
  4. Correlate their immunohistochemical expression with the demographic parameters and assess the correlation between their expression in PAS specimens.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanaa Mohammed Mohammed Sayed, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided